CLINICAL TRIAL: NCT07185360
Title: Liver Diseases: Extracellular Vesicles as Biomarkers
Acronym: LIVER-TRACK
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: APHP250409
Record Dates: First submitted 2025-08-26; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-03

CONDITIONS: Liver Diseases
Keywords: liver decompensation; extracellular vesicles; hepatocellular carcinoma; cirrhosis
MeSH Terms: conditions — Liver Diseases; Hepatic Insufficiency; Carcinoma, Hepatocellular; Fibrosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Volunteers without liver disease (Other): Volunteers without liver disease
  Interventions: Other: blood sampling for volunteers
- Diabetic patients with F3/F4 fibrosis recruited and followed prospectively (Other): Diabetic patients with F3/F4 fibrosis recruited and followed prospectively
  Interventions: Other: blood sampling for diabetics patients with F3/F4 fibrosis
- Patients with liver disease (Other): Patients with liver disease
  Interventions: Other: blood sampling for patients with liver disease

INTERVENTIONS:
Other: blood sampling for volunteers — A 38.5 ml blood sample will be taken to test for research taken to test for research
  Arms: Volunteers without liver disease
Other: blood sampling for diabetics patients with F3/F4 fibrosis — 32.5 ml will be sampled at inclusion, at one year visit and two year visit
  Arms: Diabetic patients with F3/F4 fibrosis recruited and followed prospectively
Other: blood sampling for patients with liver disease — A blood sample of 35.5 mL maximum will be taken for research purposes at the inclusion visit, M1 visit and M3 visit.
  Arms: Patients with liver disease

SUMMARY:
Worldwide, cirrhosis is responsible for 2 million deaths per year. Hepatocellular carcinoma (HCC) accounts for 800,000 of these deaths and is the 3rd leading cause of cancer related death. Cirrhosis affects mainly a working age population, hence its heavy economic burden.While patients with compensated cirrhosis do not have symptoms and have a 10-year life expectancy, decompensation of cirrhosis heralds a dramatic decrease in life expectancy to 2 years. Biomarkers allowing reliable estimation of the risk for decompensation of cirrhosis would allow community-based care, possibly by nurse practitioners, of patients at low risk, while patients had high risk could be managed in secondary and tertiary care centers and included in clinical trials. Because HCC is usually asymptomatic at early stages, when it is still curable, it can easily be missed. Biomarkers allowing stratification of the risk of HCC would allow reinforced surveillance (using magnetic resonance imaging) of high-risk patients, and their inclusion in chemoprevention clinical trials.

LIVER-TRACK aims at reliably predicting the outcome of patients with compensated cirrhosis through the development of a Tests for Decompensation and a Test for HCC. This will be achieved through leveraging circulating extracellular vesicles (EVs), an untapped source of biomarkers in liver diseases, as prognostic indicators, and combining them with existing blood biomarkers and single-nucleotide polymorphisms (SNPs). LIVER-TRACK also aims at delivering technologies for EV measurement that are useable in medical practice.

DETAILED DESCRIPTION:
Worldwide, cirrhosis is responsible for 2 million deaths per year. Hepatocellular carcinoma (HCC) accounts for 800,000 of these deaths and is the 3rd leading cause of cancer related death. Cirrhosis affects mainly a working age population, hence its heavy economic burden. While patients with compensated cirrhosis do not have symptoms and have a 10-year life expectancy, decompensation of cirrhosis heralds a dramatic decrease in life expectancy to 2 years. Biomarkers allowing reliable estimation of the risk for decompensation of cirrhosis would allow community-based care, possibly by nurse practitioners, of patients at low risk, while patients had high risk could be managed in secondary and tertiary care centers and included in clinical trials. Because HCC is usually asymptomatic at early stages, when it is still curable, it can easily be missed. Biomarkers allowing stratification of the risk of HCC would allow reinforced surveillance (using magnetic resonance imaging) of high-risk patients, and their inclusion in chemoprevention clinical trials.

LIVER-TRACK aims at reliably predicting the outcome of patients with compensated cirrhosis through the development of a Tests for Decompensation and a Test for HCC. This will be achieved through leveraging circulating extracellular vesicles (EVs), an untapped source of biomarkers in liver diseases, as prognostic indicators, and combining them with existing blood biomarkers and single-nucleotide polymorphisms (SNPs). LIVER-TRACK also aims at delivering technologies for EV measurement that are useable in medical practice.

LIVER-TRACK outputs are expected to: i) improve care for individual patients at highest medical need, i.e., patients with cirrhosis with high risk of decompensation or HCC; ii) decrease cirrhosis burden for public health, iii) facilitate drug development; and iv) technically allow exploitation of EVs as biomarkers in clinical practice, an obligatory step permitting expansion to other fields such as cancer and cardiovascular diseases.

ELIGIBILITY:
Volunteers without liver disease

- Inclusion criteria: Major

Exclusion Criteria:

* Known liver disease
* Active cancer
* Viral or bacterial infection within 2 weeks of inclusion (respiratory, dermatological, urinary, digestive, etc.)
* Transfusion in the month preceding inclusion
* Current participation or less than 3 months' participation in a therapeutic interventional trial
* Absence of signed informed consent
* Not affiliated to a social security scheme
* Pregnant women
* Person under guardianship or trusteeship

Diabetic patients with F3/F4 fibrosis recruited and followed prospectively

Inclusion criteria:

* Patient aged 18 or over
* Type 2 diabetic (ADA/WHO criteria recalled in section 20.5)
* Hepatic fibrosis stage F3/F4 on liver biopsy or hepatic elasticity > 10 kPa

Exclusion criteria:

Vulnerable person: a person deprived of liberty by a judicial or administrative decision, or under psychiatric care, and a person admitted to a health or social institution for purposes other than research.

* Protected adult
* Not affiliated to or not benefiting from a social security scheme
* Pregnant or breast-feeding women
* Absence of signed informed consent
* Illness linked to other etiologies:

  * Alcoholic liver disease
  * Current hepatitis B virus infection
  * Current hepatitis C virus infection
  * Autoimmune hepatitis according to according to AASLD and EASL recommended criteria
  * Transferrin saturation >50%
  * Alpha antitrypsin ZZ or SZ type deficiency
  * Wilson's disease
  * Liver transplant patients
  * Ultrasound obstruction of blood vessels or bile ducts (on routine ultrasound). If nothing is mentioned on the report, it is considered that there is no obstruction of the blood vessels or bile ducts).
* Current participation or less than 3 months' participation in a therapeutic interventional trial

Patients with liver disease :

Inclusion criteria:

* Major
* Child-Pugh A, B or C cirrhosis, diagnosed on the basis of histological evidence or liver elasticity > 15 kPa or a combination of biological and radiological signs.

Exclusion criteria:

* Presence of one of the following diseases in the 15 days prior to inclusion: acute renal failure, bacterial infection (proven or suspected on clinico-biological criteria), digestive bleeding,
* alcoholic hepatitis in the month prior to inclusion
* Previous porto-systemic shunt, liver transplantation, primary sclerosing cholangitis, primary biliary cholangitis, Budd-Chiari syndrome
* Active or past hepatocellular carcinoma
* Active extrahepatic neoplasia,
* Current participation or less than 3 months' participation in a therapeutic interventional trial
* Absence of signed informed consent
* Non affiliation to a social security scheme
* Pregnant or breast-feeding
* Person under guardianship or trusteeship

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 845 (Estimated)
Dates: Start 2025-09-22 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Decompensation Test in patients with cirrhosis | 48 months after the beginning of the project
  The discriminating power of the Decompensation Test will be measured using the C-index
HCC Test in patients with cirrhosis | 48 months after the beginning of the project
  The discriminating power of the HCC Test will be measured using the C-index

SECONDARY OUTCOMES:
Quantification of Extracellular vesicles proteins | 48 months after the beginning of the project
  Number of extracellular vesicles
Size of Extracellular vesicles proteins and the experimental repeatability | 48 months after the beginning of the project
  size of extracellular vesicles in nm
3D morphology of extracellular vesicles | 48 months after the beginning of the project
  size of microvesicles in nm
Extracellular vesicles plasma concentrations in the general population | 48 months after the beginning of the project
  Extracellular vesicles concentration per mL
number of patients with extreme values of extracellular vesicles in the general population | 48 months after the beginning of the project
  Extracellular vesicles concentration per mL

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Emmanuel RAUTOU, Principal Investigator — APHP
Locations (1):
- Bichat Hospital, Beaujon Hospital, Cochin Hospital and Lariboisière Hospital, Paris, France, France